CLINICAL TRIAL: NCT00557089
Title: Randomized, Placebo-controlled Trial on the Effect of rhDNase on Ventilation Inhomogeneity in Patients With Cystic Fibrosis
Brief Title: The Effect of rhDNase on Ventilation Inhomogeneity in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Felix Ratjen, Division Head, Respiratory Medicine, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000010903
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Cystic Fibrosis
Keywords: Pediatrics; Cystic Fibrosis; Lung Clearance Index; rhDNAse
MeSH Terms: conditions — Cystic Fibrosis | interventions — dornase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): This arm will receive the active treatment for 28 days, followed by a 28 day washout period and then the placebo treatment for 28 days.
  Interventions: Drug: rhDNAse; Other: Placebo
- 2 (Other): This arm will receive the placebo treatment for 28 days, followed by a 28 day washout period and then the active treatment for 28 days.
  Interventions: Drug: rhDNAse; Other: Placebo

INTERVENTIONS:
Drug: rhDNAse — 2.5 mg rhDNase will be dispensed in 2.5 ml vials and administered once a day for 28 days. Treatment will be administered by inhalation.
  Other Names: Brand Name: Pulmozyme
Other: Placebo — 2.5 mg of the placebo will be dispensed in 2.5 ml vials and administered once a day over 28 days. Treatment will be administered by inhalation.

SUMMARY:
This study will assess whether rhDNase treatment improves ventilation inhomogeneity as assessed by lung clearance index (LCI) in patients with cystic fibrosis (CF).

DETAILED DESCRIPTION:
Life expectancy in CF patients has greatly increased due to improved clinical care. While this is certainly beneficial to CF patients, it has made it more difficult to assess the effect of therapeutic interventions. Currently, FEV1 remains the primary outcome parameter for most clinical trials, but many CF patients have normal pulmonary function and the annual rate of decline is now less than 2 %. Therefore, additional parameters are needed that are more sensitive to define abnormalities in CF patients and that can be used in therapeutic trials.

Gas mixing techniques have been shown to be sensitive parameters to define abnormalities in patients with cystic fibrosis, but it is unclear how useful this technique is to detect changes after a therapeutic intervention. Abnormalities in gas clearance from the lung are largely due to retention of inhaled gases due to mucous obstruction in the lower airways and can be assessed with the lung clearance index (LCI). Interventions that improve mucous accumulation are expected to improve lung clearance as assessed by this technique. RhDNase has been demonstrated to improve lung function and reduce pulmonary exacerbations in patients with cystic fibrosis due to improved mucus clearance.

Lung clearance index (LCI) has been shown to be more sensitive than spirometry in detecting abnormalities in CF patients. Clear cut-offs have been found which can differentiate normal patients from even newly diagnosed CF patients. However, little is known about how LCI may change with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF as defined by clinical features of CF and a documented sweat chloride > 60 mEq/L by quantitative pilocarpine iontophoresis test or a genotype showing two well characterized disease causing mutations
* Informed consent and verbal assent (as appropriate) has been provided by the subject's parent or legal guardian and the subject
* 6-18 years of age at enrolment
* Able to perform reproducible spirometry
* Clinically stable at enrolment
* Ability to comply with medication use, study visits and study procedures as judged by the site investigator
* FEV1 % predicted > 70 % as calculated by the Wang reference equations

Exclusion Criteria:

* Respiratory culture positive for:

  * NTM within past year or AFB positive at screening (sputum only)
  * B. cepacia complex within past year or at screening
* Use of intravenous antibiotics or oral quinolones within 14 days of screening
* Investigational drug use within 30 days of screening
* History of alcohol, illicit drug or medication abuse within 1 year of screening
* Other major organ dysfunction excluding pancreatic dysfunction
* History of lung transplantation or currently on lung transplant list
* Physical findings at screening that would compromise the safety of the participant or the quality of the study data

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The change in LCI from baseline to end of treatment in rhDnase treated patients versus patients receiving placebo | The duration of the patient's involvement in the study (approximately 3 months)

SECONDARY OUTCOMES:
Change in FEV1 % predicted | The duration of the patient's involvement in the study (approximately 3 months)
Change in FVC (in litres) | The duration of the patient's involvement in the study (approximately 3 months)
Change in FVC % predicted | The duration of the patient's involvement in the study (approximately 3 months)
Change in FEF25-75 (liters/sec) | The duration of the patient's involvement in the study (approximately 3 months)
Change in FEF25-75 % predicted | The duration of the patient's involvement in the study (approximately 3 months)
Change in exhaled nitric oxide concentrations | The duration of the patient's involvement in the study (approximately 3 months)
Incidence of adverse events and serious adverse events | Duration of the study (approximately 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Ratjen, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Amin R, Subbarao P, Lou W, Jabar A, Balkovec S, Jensen R, Kerrigan S, Gustafsson P, Ratjen F. The effect of dornase alfa on ventilation inhomogeneity in patients with cystic fibrosis. Eur Respir J. 2011 Apr;37(4):806-12. doi: 10.1183/09031936.00072510. Epub 2010 Aug 6. PMID 20693248
- [Derived] Yang C, Montgomery M. Dornase alfa for cystic fibrosis. Cochrane Database Syst Rev. 2021 Mar 18;3(3):CD001127. doi: 10.1002/14651858.CD001127.pub5. PMID 33735508